CLINICAL TRIAL: NCT04245709
Title: A Clinical Investigation of the Safety and Efficacy of Clenbuterol on Motor Function in Individuals With Amyotrophic Lateral Sclerosis
Brief Title: Clenbuterol on Motor Function in Individuals With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dwight Koeberl, M.D., Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Dwight Koeberl, M.D., Ph.D., Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103668
Record Dates: First submitted 2020-01-26; First posted 2020-01-29 (Actual); Results first posted 2022-09-06 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Clenbuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label Arm (Experimental): This is an open label pilot trial in which 25 people with ALS will take clenbuterol orally at 40-80 micrograms twice daily for 24 weeks.
  Interventions: Drug: Clenbuterol

INTERVENTIONS:
Drug: Clenbuterol — The intervention is treatment with oral clenbuterol at 40-80 micrograms twice daily for 24 weeks. Dosage will initially be 40 mcg daily for one week, then 40 mcg BID per oral daily for the next 5 weeks. If the 40 mcg BID per oral is well tolerated in the opinion of Dr. Bedlack, the dose will be increased to 80 mcg each morning/40 mcg each evening for one week, followed by 80 mcg BID per oral for the remainder of the study. The selected target dose (80 mcg BID) is based upon the experience with the long-term administration of clenbuterol, specifically the beneficial muscle effects in a Phase I/II clinical trial that enrolled patients with late-onset Pompe disease who were previously treated with enzyme replacement therapy (Koeberl et al. 2018).

SUMMARY:
The purpose of this study is to assess the safety and tolerability of clenbuterol (taken by mouth) in subjects with ALS (amyotrophic lateral sclerosis) and to assess the effectiveness of clenbuterol with regard to motor function in subjects with ALS. Subjects will be in this study approximately 24 weeks. The study drug, clenbuterol, is taken twice a day. As part of this study subjects will have the following tests and procedures: medical history, vital signs, physical examination, blood tests, heart and lung function tests, muscle function test, ALSFRS-R (ALS Functional Rating Scale Revised), thyroid function and for women who can become pregnant, pregnancy tests.

DETAILED DESCRIPTION:
This is an open label pilot trial in which 25 people with ALS will take clenbuterol orally at 40-80 micrograms twice daily for 24 weeks. In person visits will occur at weeks 0, 4, 12 and 24. Telephone visits will occur at weeks 1, 6, 16 and 20. During these visits several safety and efficacy outcome measures will be performed for research purposes including safety labs, thyroid functions, pregnancy testing, ALSFRS-R, FVC (forced vital capacity), and muscle strength testing (myometry). The critical test of treatment efficacy will be the comparison of the ALSFRS-R slope during treatment to the estimated pre-treatment slope. All participants will continue to have standard follow up care for their ALS at Duke (for patients followed here) or their local ALS clinic

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of possible or more definite ALS according to the El Escorial criteria
* FVC >50% of predicted for age, height and gender.
* At least four of 12 ALSFRS-R questions scored as 2 or 3 at screening.
* Diminished but measurable grip strength (1) in at least one hand (females:10-50 pounds; males, 10-70 pounds).
* Taking riluzole at a stable dose or not taking riluzole at screening.
* On Radicava at a stable dose for at least 30d or not taking this
* Life expectancy at least 6 months
* Able to swallow tablets without crushing.
* Age: 18+ years at enrollment.
* Subjects are capable of giving written consent.
* If sexually active, must agree to use contraceptive or abstinence for duration of treatment
* Females of child bearing age must have negative pregnancy test at screening

Exclusion Criteria:

* Concurrent illness or laboratory abnormalities that could confound the measurement of ALS progression or interfere with the ability to complete the study.
* Taking any investigational study drug within 30 days of screening or five half-lives of the prior agent.
* No previous exposure to clenbuterol.
* Pregnancy
* Clinically relevant EKG abnormality (arrhythmia, cardiomyopathy)
* Tachycardia (resting heart rate greater than 100 beats per minute)
* History of seizure disorder
* Hyperthyroidism
* Pheochromocytoma
* Pregnancy
* Have any other co-morbid conditions that in the opinion of the study investigator, places the participant at increased risk of complications, interferes with study participation or compliance, or confounds study objectives
* History of hypersensitivity to 2-agonist drugs such as albuterol, levalbuterol (Xopenex), bitolterol (Tornalate), pirbuterol (Maxair), terbutaline, salmeterol (Serevent).
* The use of the following concomitant meds is prohibited during the study:

diuretics (furosemide, Lasix), digoxin (digitalis, Lanoxin);blockers such as atenolol (Tenormin), metoprolol (Lopressor), and propranolol (Inderal); tricyclic antidepressants such as amitriptyline (Elavil, Etrafon), doxepin (Sinequan), imipramine (Janimine, Tofranil), and nortriptyline (Pamelor); monoamine oxidase inhibitors such as isocarboxazid (Marplan), phenelzine (Nardil), rasagiline (Azilect), selegiline (Eldepryl, Emsam), or tranylcypromine (Parnate); or other bronchodilators such as albuterol (Ventolin), levalbuterol (Xopenex), bitolterol (Tornalate), pirbuterol (Maxair), terbutaline (Brethine, Bricanyl), salmeterol (Serevent), isoetherine (Bronkometer), metaproterenol (Alupent, Metaprel), or isoproterenol (Isuprel Mistometer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
there is no plan to share individual participant data (IPD) with other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label Arm
Started | 25
Completed | 11
Not Completed | 14
Not completed — Adverse Event | 13
Not completed — Risk of travel during COVID19 pandemic | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was determined as follows: Intention to treat analyses were performed for 20 participants (of 25 enrolled) who had at least one ALSFRS-R measurement post-treatment.
Groups:
- Open Label Arm: This is an open label pilot trial in which 25 people with ALS will take clenbuterol orally at 40-80 micrograms twice daily for 24 weeks.
  Clenbuterol: The intervention is treatment with oral clenbuterol at 40-80 micrograms twice daily for 24 weeks. Dosage will initially be 40 mcg daily for one week, then 40 mcg BID per oral daily for the next 5 weeks. If the 40 mcg BID per oral is well tolerated in the opinion of Dr. Bedlack, the dose will be increased to 80 mcg each morning/40 mcg each evening for one week, followed by 80 mcg BID per oral for the remainder of the study. The selected target dose (80 mcg BID) is based upon the experience with the long-term administration of clenbuterol, specifically the beneficial muscle effects in a Phase I/II clinical trial that enrolled patients with late-onset Pompe disease who were previously treated with ERT (Koeberl et al. 2018).
Arm/Group | Open Label Arm
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 59 [32 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events as Measured by Patient Reporting
Description: The primary endpoint is safety of clenbuterol at 80 mcg BID. Adverse events and serious adverse events will be systematically gathered as the dose is increased.
Time Frame: Up to 24 weeks
Population: Intention to treat analyses were performed for 20 participants who had at least one ALSFRS-R measurement post-treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Arm
Number analyzed (Participants) | 20
Participants | 2

2. Secondary Outcome: Change in Motor Function Measured by ALSFRS-R
Description: The ALS Functional Rating Scale (ALSFRS-R) - 12 questions rated on a five-point scale, where 0= can't do, to 5= normal ability. It is utilized for monitoring the progression of disability in patients with ALS. The critical test for efficacy was comparison of the mean slope of the ALSFRS-R during treatment compared to pre-treatment. Pre-treatment slope for each participant was estimated as follows: (48-enrollment ALSFRS-R)/months since symptom onset. A statistically significant treatment effect was determined by a two-tailed, t-test, with a critical p value < .05. Other analyses included a repeated measures ANOVA design (between and within subjects) of ALSFRS-R slopes before and during treatment.
Time Frame: Baseline, week 4, week 12, week 16, week 20, and week 24
Population: Intention to treat analyses were performed for 20 participants who had at least one ALSFRS-R measurement post-treatment. These calculations for ALSFRS-R were based on the 11 patients who completed all 6 months on some dose of the drug, e.g. the per-protocol group.
Measure: Mean (Standard Deviation); unit: slope
Arm/Group | Open Label Arm
Number analyzed (Participants) | 11
slope | -0.17 (0.25)

3. Secondary Outcome: FVC Decline, Per-protocol Comparison
Description: Comparison of the mean slope of percent predicted FVC during treatment versus pre-treatment. Pre-treatment slope for each participant was estimated as follows: (100%-enrollment percent predicted FVC)/months since symptom onset.
Time Frame: Baseline, week 4, week 12, and week 24
Population: For the 11 patients who completed all 6 months on some dose of the drug, there were 10 who had at least two FVC measurements. Seven patients had a baseline FVC measurement which was used to calculate the pre-treatment slope estimate, for the 3 patients without a baseline measurement, imputation of the baseline FVC was performed using all data available for each patient.
Measure: Mean (Standard Deviation); unit: slope
Arm/Group | Open Label Arm
Number analyzed (Participants) | 10
slope | -0.25 (0.85)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Open Label Arm
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Arm (N=25)
Near-drowning accident (Injury, poisoning and procedural complications) | 1 (1) — The participant was swimming and became submerged for some time before being rescued and recovering.
Pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient developed pulmonary emboli during the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Arm (N=25)
Jitters/tremors (Nervous system disorders) | 10 (10)
Insomnia (General disorders) | 7 (7)
Cramps/spasms (Musculoskeletal and connective tissue disorders) | 8 (8)
Stiffness/spasticity (Nervous system disorders) | 6 (6)
Elevated liver transaminases (Hepatobiliary disorders) | 3 (3)
Increased work of breathing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decreased appetite/weight loss (General disorders) | 2 (2)
GI upset/nausea (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Elevated creatine kinase (CK) (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Elevated PSA (Renal and urinary disorders) | 1 (1)
Tooth removal (General disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Restless legs (Nervous system disorders) | 1 (1)
Tendinitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (General disorders) | 1 (1)
Dizziness/instability (Nervous system disorders) | 1 (1)
Increased fasciculations (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
ECG changes (Cardiac disorders) | 1 (1)
Elevated thyroxine (T4) (Endocrine disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Accelerated disease progression (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT04245709/Prot_SAP_000.pdf